CLINICAL TRIAL: NCT05612581
Title: A Platform Study Evaluating the Efficacy and Safety of Investigational Therapies in Participants With Chronic Hepatitis B Infection (PREVAIL)
Brief Title: A Platform Study to Evaluate Investigational Therapies in Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-MHB1-V200
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- STRIVE: Cohort 1a (VIR-3434 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + TDF for 44 weeks total
  Interventions: Drug: VIR-3434; Drug: TDF
- STRIVE: Cohort 2a (VIR-3434 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + TDF for 44 weeks total
  Interventions: Drug: VIR-3434; Drug: TDF
- STRIVE: Cohort 3a (VIR-3434 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + TDF for 36 or 40 weeks total
  Interventions: Drug: VIR-3434; Drug: TDF
- STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + VIR-2218 + TDF for 20 or 44 weeks total
  Interventions: Drug: VIR-3434; Drug: VIR-2218; Drug: TDF
- STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) (Experimental): Participants will receive combination therapy with VIR-3434 + VIR-2218 +TDF + PEG-IFNα for 48 weeks total
  Interventions: Drug: VIR-3434; Drug: VIR-2218; Drug: TDF; Drug: PEG-IFNα
- THRIVE: Cohort 1b (VIR-3434 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + TDF for 44 weeks
  Interventions: Drug: VIR-3434; Drug: TDF
- THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF) (Experimental): Participants will receive combination therapy with VIR-3434 + VIR-2218 + TDF for 44 weeks total
  Interventions: Drug: VIR-3434; Drug: VIR-2218; Drug: TDF

INTERVENTIONS:
Drug: VIR-3434 — VIR-3434 given by subcutaneous injection
  Other Names: Tobevibart
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Other Names: Elebsiran
  Arms: STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF); STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα); THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF)
Drug: TDF — TDF given orally
Drug: PEG-IFNα — PEG-IFNα given by subcutaneous injection
  Arms: STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα)

SUMMARY:
This is a Phase 1b/2 platform study framework to evaluate the safety and efficacy of investigational candidate(s) and their combinations as potential treatments for adults with chronic hepatitis B virus infection.

DETAILED DESCRIPTION:
VIR-SHB1-V201 (STRIVE) Sub-Protocol A is a Phase 2 study under the PREVAIL platform trial. This is a multi-center, open-label study designed to evaluate the safety and efficacy of regimens containing VIR-3434, VIR-2218, PEGASYS (PEG-IFNα), and nucleotide reverse transcriptase inhibitors (NRTI) in noncirrhotic adult participants with chronic HBV infection that have not received prior NRTI or PEGASYS treatment.

VIR-SHB1-V202 (THRIVE) Sub-Protocol B is a Phase 2 study under the PREVAIL platform trial. This is a multi-center open-label study designed to evaluate the safety and efficacy of regimens containing VIR-3434 and NRTI with or without VIR-2218 in noncirrhotic adult participants with low viral burden of chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 or older
* Chronic HBV infection for >/= 6 months
* Chronic HBV infection defined as a positive serum HBsAg, HBV DNA, or HBeAg on 2 occasions at least 6 months apart based on previous or current laboratory documentation
* STRIVE: HBeAg positive or negative, HBV DNA > 2,000 IU/mL, ALT > ULN and ≤ 5x ULN
* THRIVE: Must be/have the following, within the 1-year period prior to screening: HBeAg negative, HBV DNA ≤ 2,000 IU/mL, ALT ≤ ULN

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the participant unsuitable for participation
* History of clinically significant liver disease from non-HBV etiology
* History or current evidence of hepatic decompensation
* Co-infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or hepatitis E virus (HEV).
* History or clinical evidence of alcohol or drug abuse
* STRIVE and THRIVE: Significant fibrosis or cirrhosis
* STRIVE and THRIVE: History of immune complex disease
* STRIVE and THRIVE: History of autoimmune disorder
* STRIVE and THRIVE: History of allergic reactions, hypersensitivity, or intolerance to monoclonal antibodies, antibody fragments, or any excipients of VIR-3434
* STRIVE: Prior NRTI or PEG-IFN therapy
* STRIVE: History of known contraindication to any interferon product
* THRIVE: Prior NRTI therapy < 24 weeks of study or any prior PEG-IFN therapy

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- France (4):
  - Investigative Site, Clichy
  - Investigative Site, Nice
  - Investigative Site, Rennes
  - Investigative Site, Toulouse
- Hong Kong (2):
  - Investigative Site, Hong Kong, Sha Tin
  - Investigative Site, Hong Kong
- Investigative Site, Chisinau, Moldova
- Investigative Site, Bucharest, Romania
- South Korea (3):
  - Investigative Site, Busan
  - Investigative Site, Seoul
  - Investigative Site, Yangsan
- United Kingdom (3):
  - Investigative Site, Glasgow
  - Investigative Site, London
  - Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not enrolled in Cohort 1a, 2a,3a, 5a and 1b Arms/Groups
Period: Overall Study
Arm/Group | STRIVE: Cohort 1a (VIR-3434 + TDF) | STRIVE: Cohort 2a (VIR-3434 + TDF) | STRIVE: Cohort 3a (VIR-3434 + TDF) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) | THRIVE: Cohort 1b (VIR-3434 + TDF) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF)
Started | 0 | 0 | 0 | 16 | 0 | 0 | 17
Completed | 0 | 0 | 0 | 11 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: cohort 1a, 2a,3a, 5a and 1b were not open for enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | STRIVE: Cohort 1a (VIR-3434 + TDF) | STRIVE: Cohort 2a (VIR-3434 + TDF) | STRIVE: Cohort 3a (VIR-3434 + TDF) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) | THRIVE: Cohort 1b (VIR-3434 + TDF) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 16 | 0 | 0 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 16 | 0 | 0 | 17 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  STRIVE: Cohort 4a |  |  |  | 43.3 (9.67) |  |  | 0 (0) | 43.3 (9.67)
  THRIVE: Cohort 2b |  |  |  | 0 (0) |  |  | 48.4 (9.78) | 48.4 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  | 10 |  |  | 9 | 19
  Male |  |  |  | 6 |  |  | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  |  | 0 |  |  | 0 | 0
  Not Hispanic or Latino |  |  |  | 16 |  |  | 17 | 33
  Unknown or Not Reported |  |  |  | 0 |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  | 0 |  |  | 0 | 0
  Asian |  |  |  | 6 |  |  | 7 | 13
  Native Hawaiian or Other Pacific Islander |  |  |  | 0 |  |  | 0 | 0
  Black or African American |  |  |  | 2 |  |  | 5 | 7
  White |  |  |  | 7 |  |  | 5 | 12
  More than one race |  |  |  | 0 |  |  | 0 | 0
  Unknown or Not Reported |  |  |  | 1 |  |  | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand |  |  |  | 0 |  |  | 0 | 0
  South Korea |  |  |  | 1 |  |  | 5 | 6
  Romania |  |  |  | 6 |  |  | 2 | 8
  Hong Kong |  |  |  | 4 |  |  | 2 | 6
  United Kingdom |  |  |  | 3 |  |  | 3 | 6
  Moldova |  |  |  | 0 |  |  | 2 | 2
  France |  |  |  | 2 |  |  | 3 | 5
  Thailand |  |  |  | 0 |  |  | 0 | 0
Hepatitis B surface antigen (Log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL]
  STRIVE: Cohort 4a |  |  |  | 3.64 (0.72) |  |  | 0 (0) | 3.64 (0.72)
  THRIVE: Cohort 2b |  |  |  | 0 (0) |  |  | 3.12 (0.66) | 3.12 (0.66)
Hepatitis B e antigen status [Count of Participants; unit: Participants]
  HBeAg positive |  |  |  | 3 |  |  | 0 | 3
  HBeAg negative |  |  |  | 13 |  |  | 17 | 30
Alanine Aminotransferase (U/L) [Mean (Standard Deviation); unit: U/L]
  STRIVE: Cohort 4a |  |  |  | 50.4 (33.26) |  |  | 0 (0) | 50.4 (33.26)
  THRIVE: Cohort 2b |  |  |  | 0 (0) |  |  | 25.3 (20.61) | 25.3 (20.61)
Hepatitis B Virus DNA (Log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL]
  STRIVE: Cohort 4a |  |  |  | 5.21 (1.71) |  |  | 0 (0) | 5.21 (1.71)
  THRIVE: Cohort 2b |  |  |  | 0 (0) |  |  | 2.61 (0.70) | 2.61 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: STRIVE and THRIVE: Proportion of Participants Achieving Suppression of HBV DNA (< LLOQ) With HBsAg Loss (< 0.05 IU/mL) at the End of Treatment
Time Frame: Up to 48 weeks
Population: Cohort 1a, 2a, 3a,5a and 1b was not opened for enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | STRIVE: Cohort 1a (VIR-3434 + TDF) | STRIVE: Cohort 2a (VIR-3434 + TDF) | STRIVE: Cohort 3a (VIR-3434 + TDF) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) | THRIVE: Cohort 1b (VIR-3434 + TDF) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF)
Number analyzed (Participants) | 0 | 0 | 0 | 16 | 0 | 0 | 17
Participants |  |  |  | 1 |  |  | 4

2. Secondary Outcome: STRIVE and THRIVE: Proportion of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

3. Secondary Outcome: STRIVE and THRIVE: Proportion of Participants With Serum HBsAg ≤ 10 IU/mL at End of Treatment
Time Frame: Up to 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: STRIVE and THRIVE: Proportion of Participants With Serum HBsAg ≤ 10 IU/mL at 24 Weeks Post-end of Treatment
Time Frame: Up to 72 weeks
Reporting Status: Not Posted

5. Secondary Outcome: STRIVE and THRIVE: Serum HBsAg Levels and Change From Baseline Across Timepoints in the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

6. Secondary Outcome: STRIVE and THRIVE: Serum HBsAg Level at Nadir During the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

7. Secondary Outcome: STRIVE and THRIVE: Time to Achieve Nadir of Serum HBsAg During the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

8. Secondary Outcome: STRIVE and THRIVE: Time to Achieve Serum HBsAg Loss (< 0.05 IU/mL)
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

9. Secondary Outcome: STRIVE and THRIVE: Proportion of Participants With HBsAg Loss With Anti-HBs Seroconversion at End of Treatment and at 24 Weeks Post-end of Treatment
Time Frame: Up to 76 weeks
Reporting Status: Not Posted

10. Secondary Outcome: STRIVE: Proportion of Participants Achieving Sustained Suppression of HBV DNA (< LLOQ) With HBsAg Loss (< 0.05 IU/mL) After Discontinuation of All Treatment at 24 Weeks and at the F48 Follow-Up Visit
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

11. Secondary Outcome: STRIVE: Proportion of Participants With HBsAg Loss (<0.05 IU/mL) at End of Treatment and at 24 Weeks Post-end of Treatment
Time Frame: Up to 72 weeks
Reporting Status: Not Posted

12. Secondary Outcome: STRIVE: Proportion of Participants Achieving Sustained Suppression of HBV DNA (< LLOQ) After Discontinuation of All Treatment at 24 Weeks and at the F48 Follow-Up Visit
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

13. Secondary Outcome: STRIVE: For HBeAg-positive Participants: Proportion of Participants With HBeAg Loss (Undetectable HBeAg) and/or Anti-HBe Seroconversion
Time Frame: Up to 72 weeks
Reporting Status: Not Posted

14. Secondary Outcome: STRIVE: Incidence and Titers of Anti-drug Antibodies (ADA; if Applicable) to VIR-3434
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

15. Secondary Outcome: STRIVE: Mean Change in Serum HBsAg Level From Baseline Across Timepoints in the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

16. Secondary Outcome: STRIVE: Proportion of Participants Achieving HBV DNA (< LLOQ) Across Timepoints in the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

17. Secondary Outcome: STRIVE: Proportion of Participants Achieving ALT ≤ ULN Across Timepoints in the Study
Time Frame: Up to 96 weeks
Reporting Status: Not Posted

18. Secondary Outcome: THRIVE: Proportion of Participants Achieving Sustained Suppression of HBV DNA (< LLOQ) With HBsAg Loss (< 0.05 IU/mL) After Discontinuation of All Treatment at 24 Weeks and at 48 Weeks
Time Frame: Up to 92 weeks
Reporting Status: Not Posted

19. Secondary Outcome: THRIVE: Proportion of Participants Achieving HBsAg Loss (< 0.05 IU/mL) at End of Treatment and at 24 Weeks Post-end of Treatment
Time Frame: Up to 44 weeks
Reporting Status: Not Posted

20. Secondary Outcome: THRIVE: Proportion of Participants Achieving Sustained Suppression of HBV DNA (< LLOQ) After Discontinuation of All Treatment at 24 Weeks and at 48 Weeks
Time Frame: Up to 68 weeks
Reporting Status: Not Posted

21. Secondary Outcome: THRIVE: Incidence and Titers of ADA (if Applicable) to VIR-3434
Time Frame: Up to 92 weeks
Reporting Status: Not Posted

22. Secondary Outcome: THRIVE: Mean Change in Serum HBsAg Level From Baseline Across Timepoints in the Study
Time Frame: Up to 92 weeks
Reporting Status: Not Posted

23. Secondary Outcome: THRIVE: Proportion of Participants Achieving HBV DNA (< LLOQ)
Time Frame: Up to 92 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 Weeks
Description: Data reported at only through primary end point collection date and final study adverse events data will be reported with final results
Arm/Group | STRIVE: Cohort 1a (VIR-3434 + TDF) | STRIVE: Cohort 2a (VIR-3434 + TDF) | STRIVE: Cohort 3a (VIR-3434 + TDF) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) | THRIVE: Cohort 1b (VIR-3434 + TDF) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/16 | 0/0 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/16 | 0/0 | 0/0 | 1/17
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 11/16 | 0/0 | 0/0 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STRIVE: Cohort 1a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 2a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 3a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) (N=16) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) (N=0) | THRIVE: Cohort 1b (VIR-3434 + TDF) (N=0) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF) (N=17)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.25% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STRIVE: Cohort 1a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 2a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 3a (VIR-3434 + TDF) (N=0) | STRIVE: Cohort 4a (VIR-3434 + VIR-2218 + TDF) (N=16) | STRIVE: Cohort 5a (VIR-3434 + VIR-2218 + TDF + PEG-IFNα) (N=0) | THRIVE: Cohort 1b (VIR-3434 + TDF) (N=0) | THRIVE: Cohort 2b (VIR-3434 + VIR-2218 + TDF) (N=17)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | NA | NA | 4
Chills (General disorders) | NA | NA | NA | 2 | NA | NA | 2
Fatigue (General disorders) | NA | NA | NA | 2 | NA | NA | 2
Pyrexia (General disorders) | NA | NA | NA | 1 | NA | NA | 2
Feeling of body temperature change (General disorders) | NA | NA | NA | 0 | NA | NA | 1
Injection site erythema (General disorders) | NA | NA | NA | 2 | NA | NA | 1
Injection site mass (General disorders) | NA | NA | NA | 0 | NA | NA | 1
Injection site paraesthesia (General disorders) | NA | NA | NA | 0 | NA | NA | 1
Pain (General disorders) | NA | NA | NA | 0 | NA | NA | 1
Injection site pain (General disorders) | NA | NA | NA | 2 | NA | NA | 0
Immediate post-injection reaction (General disorders) | NA | NA | NA | 1 | NA | NA | 0
Injection site oedema (General disorders) | NA | NA | NA | 1 | NA | NA | 0
Injection site pruritus (General disorders) | NA | NA | NA | 1 | NA | NA | 0
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 2 | NA | NA | 2
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | NA | NA | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | NA | NA | 1
COVID-19 (Infections and infestations) | NA | NA | NA | 1 | NA | NA | 1
Pharyngitis (Infections and infestations) | NA | NA | NA | 0 | NA | NA | 1
Upper respiratory tract infection (Infections and infestations) | NA | NA | NA | 2 | NA | NA | 1
Tracheitis (Infections and infestations) | NA | NA | NA | 1 | NA | NA | 0
Conjunctivitis allergic (Eye disorders) | NA | NA | NA | 0 | NA | NA | 1
Vision blurred (Eye disorders) | NA | NA | NA | 0 | NA | NA | 1
Excessive eye blinking (Eye disorders) | NA | NA | NA | 1 | NA | NA | 0
Abdominal distension (Gastrointestinal disorders) | NA | NA | NA | 0 | NA | NA | 1
Abdominal pain (Gastrointestinal disorders) | NA | NA | NA | 0 | NA | NA | 1
Gastritis (Gastrointestinal disorders) | NA | NA | NA | 0 | NA | NA | 1
Nausea (Gastrointestinal disorders) | NA | NA | NA | 2 | NA | NA | 1
Vomiting (Gastrointestinal disorders) | NA | NA | NA | 2 | NA | NA | 1
Abdominal discomfort (Gastrointestinal disorders) | NA | NA | NA | 1 | NA | NA | 0
Rectal haemorrhage (Gastrointestinal disorders) | NA | NA | NA | 1 | NA | NA | 0
Headache (Nervous system disorders) | NA | NA | NA | 5 | NA | NA | 2
Tension headache (Nervous system disorders) | NA | NA | NA | 1 | NA | NA | 0
Cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 2 | NA | NA | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | NA | NA | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | NA | NA | 1
Hypertension (Vascular disorders) | NA | NA | NA | 0 | NA | NA | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | NA | NA | NA | 0 | NA | NA | 1
Neutropenia (Blood and lymphatic system disorders) | NA | NA | NA | 1 | NA | NA | 1
Hepatic cyst (Hepatobiliary disorders) | NA | NA | NA | 0 | NA | NA | 1
Ligament sprain (Injury, poisoning and procedural complications) | NA | NA | NA | 0 | NA | NA | 1
Alpha 1 foetoprotein increased (Investigations) | NA | NA | NA | 3 | NA | NA | 0
Alanine aminotransferase increased (Investigations) | NA | NA | NA | 0 | NA | NA | 1
Aspartate aminotransferase increased (Investigations) | NA | NA | NA | 0 | NA | NA | 1
Blood creatine phosphokinase increased (Investigations) | NA | NA | NA | 0 | NA | NA | 1
Ovarian cyst (Reproductive system and breast disorders) | NA | NA | NA | 0 | NA | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may present or publish results after:

* the study results in their entirety have been publicly disclosed by or with the consent of the Sponsor OR study has been completed at all investigative sites for at least 2 years.
* provision of publication 90 days before planned submission to allow Sponsor to remove confidential information or identify Sponsor intellectual property Publication may be delayed as applicable up to 6 months for Sponsor to file patent application(s)

DOCUMENTS (4):
  • Study Protocol: PREVAIL (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT05612581/Prot_000.pdf
  • Study Protocol: STRIVE (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT05612581/Prot_001.pdf
  • Study Protocol: THRIVE (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT05612581/Prot_002.pdf
  • Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05612581/SAP_003.pdf